CLINICAL TRIAL: NCT00111215
Title: Treatment and Management of Women With Bleeding Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCBDDD-2906
Record Dates: First submitted 2005-05-18; First posted 2005-05-19 (Estimated); Last update posted 2007-03-13 (Estimated); Status verified 2006-06

CONDITIONS: Menorrhagia; Blood Coagulation Disorders; Blood Platelet Disorders; Von Willebrand Disease; Hematologic Disease
Keywords: Menorrhagia; Von Willebrand's Disease; Platelet Disorder
MeSH Terms: conditions — Menorrhagia; Blood Coagulation Disorders; Blood Platelet Disorders; von Willebrand Diseases; Hematologic Diseases | interventions — Tranexamic Acid; Deamino Arginine Vasopressin

INTERVENTIONS:
Drug: Tranexamic Acid
Drug: Desmopressin Acetate

SUMMARY:
The purpose of the study is to determine whether oral contraceptives, desmopressin acetate, and/or tranexamic acid are effective in the treatment of women with menorrhagia who are diagnosed with a bleeding disorder.

DETAILED DESCRIPTION:
Menorrhagia is a common clinical problem. Morbid events include dysmenorrhea, hospitalizations, red blood cell transfusions, and quality of life impairment in terms of daily activities, chronic pain, and time lost from work and or school. Up to 60% of women with uncontrolled menorrhagia undergo hysterectomy. Up to 20% of women with menorrhagia may have undiagnosed von Willebrand disease (vWd), or other bleeding disorders. Prevalence of vWd in the general population is estimated at just over 1%. Intuitively, the prevalence of vWd in women with menorrhagia is probably higher since platelet plug formation is necessary for menstrual hemostasis. Current management of menorrhagia in patients in the United States often begins with hormonal therapy. Estrogen and estrogen derivatives in oral contraceptives have been shown to increase von Willebrand factor (vWf) levels. Women with menorrhagia who have vWd or who are hemophilia A carriers have also been successfully treated with desmopressin acetate (DDAVP, Stimate® Nasal Spray). Tranexamic acid (Cyklokapron) is utilized extensively for menorrhagia in Australia and the United Kingdom. Standard hormonal therapy has not been compared with desmopressin or antifibrinolytics for menorrhagia. This study will compare treatment options for women with menorrhagia who have a detectable bleeding disorder. Investigators will document the effect on quality of life, menstrual flow, and coagulation parameters of treatment with oral contraceptive pills, desmopressin, or tranexamic acid.

ELIGIBILITY:
Inclusion Criteria:

* Referred to study by gynecologist or internist/family practitioner with diagnosis of menorrhagia or referred by self through community advertising or networking
* Prospective pictorial chart scores of menses >100
* Negative pelvic exam and Pap smear within the past year. *Ultrasound if manual exam indicates abnormal uterine size; *Endometrial biopsy if >35 and non-cyclic bleeding; *Rule out acute pelvic diseases - gonorrhea, chlamydia
* Age 18-50
* Willing to go off oral contraceptives and selected drugs (including some nutritional supplements and drugs that affect coagulation such as aspirin and ibuprofen) for initial laboratory testing and throughout the cross-over drug portion of the study
* Periods at least every 39 days

Exclusion Criteria:

* Patient is not proficient in English
* Patient is pregnant
* Patient on hormone replacement, Depo-Provera, or Norplant in last three months
* Patient has intrauterine device (IUD) present
* Patient is taking warfarin sodium (Coumadin) or other anti-coagulation therapy
* History of documented vascular disease (coronary artery disease, cerebrovascular disease or stroke, transient ischemic attack, peripheral vascular disease)
* Uncontrolled hypertension
* Insulin dependent diabetes mellitus
* Chronic renal or liver disease
* History of seizure disorder
* History of cancer (other than non-invasive skin cancer)
* History of venous or arterial thromboembolism
* Patient with a previously diagnosed bleeding disorder has taken or is taking desmopressin acetate or antifibrinolytic drugs for treatment of heavy menstrual bleeding

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100
Dates: Start 2001-01; Study Completion 2006-09

PRIMARY OUTCOMES:
Reduction of menstrual blood loss as measured by a Pictorial Self-Assessment Chart
Changes in quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Nicole F Dowling, PhD, Study Director — Centers for Disease Control and Prevention
Locations (6):
- United States (6):
  - Emory University School of Medicine, Atlanta, Georgia
  - Michigan State University, East Lansing, Michigan
  - The Mayo Clinic, Rochester, Minnesota
  - UMDNJ Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Mary M. Gooley Hemophilia Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina